CLINICAL TRIAL: NCT06277583
Title: Effects of Urban Care Farming on Promoting Wellbeing and Productive Engagement for Older Adults: A Randomised Controlled Trial
Brief Title: Urban Care Farming on Living Well and Productive Engagement of Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Chen Huijun, Cynthia, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NUS-IRB-2023-191
Record Dates: First submitted 2023-12-01; First posted 2024-02-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2024-02

CONDITIONS: Stress, Psychological
Keywords: stress; quality of life; biopsychosocial
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Waitlist controlled trials: Participants from both the intervention and waitlist control groups will undergo the intervention 6 months apart.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urban Care farming Intervention (Experimental): This intervention group of participants will receive the experimental urban care farming treatment.
  Interventions: Behavioral: Urban care farming
- Waitlist control (Other): Waitlist control group consists of participants who do not receive the experimental treatment, but who are put on a waiting list to receive the intervention after the active treatment group does.
  Interventions: Behavioral: Urban care farming

INTERVENTIONS:
Behavioral: Urban care farming — An intervention curriculum has been designed using horticulture therapy combined with urban farming techniques. The sessions will use plants and interaction with nature to engage and rehabilitate participants. Both the intervention and control group participants will undergo the intervention. But the intervention group will start with the urban care farming intervention first, and the control group will follow once the intervention group completes the program.

SUMMARY:
The goal of the randomized controlled trials is to learn about the effects of urban farming interventions on older adults' physical, mental, and social well-being of older adults aged 50 to 85 years. The main questions the study aims to answer are Q1. Would participants who have undergone the urban care farming intervention have lower stress levels compared to those who did not undergo the intervention? Q2. Would the quality of life and biopsychosocial factors of older adults who participate in the urban farming interventions be better before the intervention and compared to those who did not participate? Q3. Would running intervention programs as such demonstrate cost-effectiveness? Participants will be enrolled in 24 weekly lessons providing hands-on urban farming techniques, including physical activity, planting, and social interactions. Researchers will compare older participants with similar demographic profile to determine if the biological, psychological, and social factors are better for the intervention group.

DETAILED DESCRIPTION:
The data collection consists of three sessions, before and after the 24-week intervention program, and 6 months post-intervention. Prior to the data collection, participants will be assessed for eligibility criteria and explained the detailed study procedures by trained research staff for informed consent. After completing the written informed consent, participants will be interviewed using detailed questionnaires relating to their health, nutrition, and dietary status, psychosocial measures, and undergo a series of physical examinations. These examinations include physical performance tests of mobility and gait, balance and strength, body measurements of weight, height, body mass index (BMI), waist-hip circumference, mid-upper-arm and calf circumference, blood pressure, and blood tests that will examine participants' clinical profile, biomarkers, and immunoassays. Participants will also be given Fitbit trackers to determine if they have improved their physical activity. Last, data collected will also include Functional near-infrared spectroscopy (fNIRS), a non-invasive procedure to determine the oxygenation levels of participants at rest and while doing some thinking activities. This data collection procedure will be conducted at baseline before the intervention and after the completion of the intervention.

The intervention will include a weekly, 24-week urban farming program. Each weekly session is where participants will engage in outdoor and indoor horticultural activities ranging from fertilization, sowing, and watering, to transplanting, maintaining, and harvesting vegetables and herbs.

ELIGIBILITY:
Inclusion Criteria:

* Willing to take part in the intervention
* Agree for their data to be used for research purposes
* Ambulant and able to carry out some tasks independently

Exclusion Criteria:

* Not willing to participate in the data collection (participants can opt not to answer some questions in the questionnaire but have to consent to the other data collection methods, e.g., Blood taking/test)
* Refusal to give informed consent
* Unable to give consent independently
* Have a disability of the upper or lower body that limits their mobility
* Have medical conditions which in the opinion of the research/investigative team that would compromise (or interfere with) their ability to participate in the study
* Had a recent severe medical episode (e.g., heart attack)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
WHO Quality of Life Scale (WHOQOL-BREF) | Baseline, 6 months, 12 months
  Brief version consisting of 26 QOL related questions developed by World Health Organisation. There are four domains, Physical, Psychological, Social relationships, and Environment. The minimum and maximum for each domain is 0 and 100 respectively, with higher scores being better outcome for each domain.

SECONDARY OUTCOMES:
Immuno-biomarkers: IL-1RA, IL-6, IL-8 (CXCL8), IL-10, IL-13, IL-17A (CTLA-8), MIP-3 beta (CCL19), SDF-1 alpha, MMP-3, MMP-9, MCP-1 (CCL2), and TNF alpha | Baseline, 6 months
  changes in concentration of cytokines, chemokines and selected ageing and inflammatory markers in measured in pg/mL
Brief sense of community scale (BSCS) | Baseline, 6 months, 12 months
  8-items measuring the dimensions of needs fulfillment, group membership, influence, and emotional connection. Composite scores with the average of the 8 items is computed, min 1 and max. 8, with higher scores showing greater sense of community.
Fried phenotype of frailty | Baseline, 6 months, 12 months
  Fried frailty phenotype (FP) assesses physical frailty through five criteria: unintentional weight loss; weakness or poor handgrip strength; self-reported exhaustion; slow walking speed; and low physical activity. Total scores are classified into 3 categories: non-frail, pre-frail, and frail.
Lubben social network scale (LSNS-6) | Baseline, 6 months, 12 months
  This scale measure of social engagement including family and friends, min score of 6 and max. score of 30. A higher score indicating more social engagement and a cutoff of 12 points indicate risk of social isolation.
Functional near-infrared spectroscopy | Baseline, 6 months
  Brain oxygenation levels measured in cerebral metabolic rate of oxygen (CMRO^2).
EQ5D | Baseline, 6 months, 12 months
  EQ5D-5L, a measure that consists five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. An utility score can be attached to the total score to determine the cost utility of the participants' quality of life. An utility score between 0 to 1 on the Singapore population will be derived.
MOCA | Baseline, 6 months, 12 months
  Participants are scored following MOCA scoring criteria. Max. 30 points. Scores lower than 26 showed signs of cognitive impairment.
Brief resilience scale | Baseline, 6 months, 12 months
  Resilience scale on a 5 points scale, strongly disagree to strongly agree, the higher the score, the greater resilience.
De jong Gierveld loneliness scale | Baseline, 6 months, 12 months
  Measures emotional and/or social loneliness situation of respondents and adds up to a total loneliness score. the total loneliness score can be categorized into four levels: not lonely (score 0, 1 or 2), moderate lonely (score 3 through 8), severe lonely (score 9 or 10), and very severe lonely (score 11).
Fitbit | Continuous for 30 weeks
  Steps count
Body weight and height | Baseline, 6 months, 12 months
  Measured in kilograms and metres respectively. Weight and height will be combined to report BMI in kg/m^2
Fasting plasma glucose, HbA1c | Baseline, 6 months
  measures average blood sugar levels over the past 3 months
Serum Creatinine | Baseline, 6 months
  measures the level of creatinine in the blood
Attitude towards eating healthy food | Baseline, 6 months, 12 months
  Attitude of healthy eating (11-items) adapted from Saba et al 2019 (DOI: 10.1016/j.foodqual.2018.11.017). Composite score computed from the averaged measures will have a min of 1 and max of 5.
Waist and hip circumference | Baseline, 6 months, 12 months
  Measured in centimetres
Blood pressure | Baseline, 6 months, 12 months
  Measured in systolic and diastolic
Lipid panel | Baseline, 6 months
  A lipid panel measures levels of various types of lipids (fats) in the blood. Measures HDL cholesterol (High-Density Lipoprotein) and LDL cholesterol (Low-Density Lipoprotein) and Triglycerides
Eating fruits and vegetables behavior | Baseline, 6 months, 12 months
  Behavior (8-items) towards eating fruits and vegetables developed for this study. Max. score of 10 and minimum score of 2 will be derived from this measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Chen, PhD, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - NUS, Singapore, Singapore
  - Jurong Lake Garden, Singapore

IPD SHARING:
Plan to Share IPD: Yes
There is plan to share data dictionaries and unidentified IPD will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: June 2024
Access Criteria: Study protocol will be published as a journal article.